CLINICAL TRIAL: NCT02992106
Title: Evolution of Maternal Weight During Pregnancy and Influence on the Endothelial Function in Her Offspring
Acronym: EFFECTOR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Collaborators: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Inge Gies, Pediatric Endocrinologist, Universitair Ziekenhuis Brussel
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: EFFECTOR
Record Dates: First submitted 2016-12-05; First posted 2016-12-14 (Estimated); Last update posted 2019-08-07 (Actual); Status verified 2019-08

CONDITIONS: Endothelial Dysfunction; Childhood Obesity
Keywords: Maternal Obesity; Endothelial Dysfunction; Childhood Obesity
MeSH Terms: conditions — Pediatric Obesity; Pregnancy in Obesity | interventions — Blood Specimen Collection; High-Energy Shock Waves

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Normal weight during pregnancy (Other): Offspring of 156 women with a normal weight during their pregnancy recruited by Bogaerts et al, in 3 belgian hospitals. Results of maternal data published in 2013. Now the children will be recruited. This group wil function as a control group.
  All participating children will undergo the same examinations:
  * Parental questionnaires
  * Blood sample
  * Urine sample
  * Anthropometric measurements
  * Abdominal ultrasound (fat mass)
  * EndoPAT
  Interventions: Other: Parental questionnaires; Other: Blood sample; Other: Urine sample; Other: Anthropometric measurements; Other: Ultrasound; Other: EndoPAT; Other: Faces Pain Scale
- Obese mothers without intervention (Other): This subgroup will be compiled of the offspring of women recruited in two different studies. First of all there is the offspring of 65 women from the cohort that was recruited by Guelinckx et al, data published in 2010. This population was recruited in the University hospital of Leuven as control group for women receiving lifestyle interventions during pregnancy. Secondly there are children of 63 women from the cohort of Bogaerts et al of 2013 that had a BMI > 29 kg/m² during their singleton pregnancy.
  All participating children will undergo the same examinations:
  * Parental questionnaires
  * Blood sample
  * Urine sample
  * Anthropometric measurements
  * Abdominal ultrasound (fat mass)
  * EndoPAT
  Interventions: Other: Parental questionnaires; Other: Blood sample; Other: Urine sample; Other: Anthropometric measurements; Other: Ultrasound; Other: EndoPAT; Other: Faces Pain Scale
- Obese mothers & lifestyle intervention (Other): This one will also be a composition of study subjects of two different study cohorts. Firstly there are children of about 100 Belgian women that were included in the DALI cohort, a European randomized controlled trial. All of them underwent a lifestyle intervention during pregnancy, concerning diet and/ or exercise. Secondly there is the offspring of the other subgroup of the cohort recruited by Guelinckx et al. 130 women were divided into 2 groups which underwent lifestyle interventions during pregnancy.
  All participating children will undergo the same examinations:
  * Parental questionnaires
  * Blood sample
  * Urine sample
  * Anthropometric measurements
  * Abdominal ultrasound (fat mass)
  * EndoPAT
  Interventions: Other: Parental questionnaires; Other: Blood sample; Other: Urine sample; Other: Anthropometric measurements; Other: Ultrasound; Other: EndoPAT; Other: Faces Pain Scale
- History of bariatric surgery (Other): The PABAS cohort (Pregnancy After Bariatric Surgery) provides children of 49 women who underwent bariatric surgery before their singleton pregnancy. The women were included in five Flemish hospitals before 15 weeks of pregnancy. Furthermore we will recruit the offspring of 200 women that are recruited in the ongoing AURORA cohort (bAriatric sUrgery Registration in women Of Reproductive Age). Women in this cohort are recruited from the start of their process undergoing bariatric surgery and are followed until after their pregnancy.
  All participating children will undergo the same examinations:
  * Parental questionnaires
  * Blood sample
  * Urine sample
  * Anthropometric measurements
  * Abdominal ultrasound (fat mass)
  * EndoPAT
  Interventions: Other: Parental questionnaires; Other: Blood sample; Other: Urine sample; Other: Anthropometric measurements; Other: Ultrasound; Other: EndoPAT; Other: Faces Pain Scale

INTERVENTIONS:
Other: Parental questionnaires — We will provide parents with questionnaires depending on the age of their children:
  * Children aged 0-6 years old:
    1. Questionnaire on socio-demographic characteristics
    2. Dutch Eating Behaviour Questionnaire
    3. Food Frequency Questionnaire
    4. Ages and Stages Questionnaire
    5. Strengths and Difficulties Questionnaire
    6. Questionnaire on developmental milestones
    7. Questionnaire on behaviour
  * Children older than 6 years:
    1. Questionnaire on socio-demographic characteristics
    2. Dutch Eating Behaviour Questionnaire
    3. Food Frequency Questionnaire
    4. Pediatric Quality of Life Questionnaire
    5. Children's Behaviour Questionnaire in Dutch
    6. Questionnaire on developmental milestones
    7. Developmental Coordination Disorder Questionnaire
    8. Strengths and Difficulties Questionnaire
Other: Blood sample — We will determine the following biochemical parameters: glucose, insulin, total cholesterol, LDL, HDL, triglycerides, uric acid, IGF-1, adiponectin, leptin, hs-CRP, IL-6, TNF-α and ICAM-1.
Other: Urine sample — We will take a urine sample to evaluate the albumin to creatinin ratio.
Other: Anthropometric measurements — We will measure weight, Height, hip, waist and neck circumference, blood pressure, 4-site skinfold measurements and BIA.
Other: Ultrasound — We will do an abdominal ultrasound to measure the abdominal fat accumulation
Other: EndoPAT — We will use the EndoPAT device to measure endothelial function, which is a non-invasive and innovative technique (peripheral pulse wave amplitude measurement).
Other: Faces Pain Scale — After performing the measurements with the EndoPAT device, Harpender kalliper and ultrasound, the children will be asked to fill out a Faces Pain Scale, validated for children aged 4-16 years old and obtained for use from the International Association for the Study of Pain

SUMMARY:
The rising worldwide prevalence of obesity and its subsequently rising incidence of concommitant diseases as diabetes and cardiovascular events impose a defiant obstacle for the health care and associated health care costs of future generations. Obese pregnant women are a growing population of interest because their offspring is at risk for childhood obesity, an adverse metabolic and inflammatory profile and possible endothelial dysfunction. However, strong evidence is still lacking regarding the hypotheses on the early origin of these long-term health consequences.

Consequently there is no comprehensive data available on the contribution of changing maternal weight through lifestyle interventions or bariatric surgery and an eventual adverse metabolic and endothelial programming of the offspring.

The investigators of this study want to provide additional data on the body composition, metabolic and inflammatory state as well as endothelial function of children of obese pregnant women women and compare the outcome with children born from normal weight women. Furthermore, the investigators of this study will stratify the obese pregnant women into 3 groups: women who did not underwent an intervention, women who underwent a weight changing intervention during pregnancy e.g. diet or lifestyle intervention and women who underwent bariatric surgery before pregnancy. The overall aim of the study is to prove that in all the diverse groups of participating children, except the control group, there will be a certain grade of endothelial dysfunction, even if there was a normalization of weight, insulin sensitivity and inflammation before conception or delivery in the mother.

ELIGIBILITY:
Inclusion Criteria:

* Children of women who previously participated in different cohort studies conducted in Flanders concerning maternal obesity are included after contacting the mothers again. During the initial clinical trials the mothers were informed of possible follow-up studies on their offspring.

Exclusion Criteria:

* There are no absolute exclusion criteria formulated.
* For the peripheral pulse wave amplitude measurement we exclude children on growth hormone therapy.
* We postpone the examination for 2 weeks if there is an ongoing infection.
* We document the use of specific medication, but the use of it doesn't implicate exclusion of the participating children.

Ages: 6 Months to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 143 (Actual)
Dates: Start 2017-05-10 (Actual); Primary Completion 2019-03-18 (Actual); Study Completion 2019-03-18 (Actual)

PRIMARY OUTCOMES:
Reactive Hyperemia Index (EndoPAT) | Through study completion, average of 18 months
  Reactive Hyperemia Index is one of the outcome parameters of the EndoPAT assessment of endothelial cell function
Albumin to creatinin ratio in urine | Through study completion, average of 18 months
  Albumin to creatinin ratio is considered an early marker of endothelial cell dysfunction
Peak response after occlusion (EndoPAT) | Through study completion, average of 18 months
  Determination of the peak response using 30s average of amplitude intervals./ In children considered as an important measurement regarding assessment of the endothelial cell function

SECONDARY OUTCOMES:
BMI (kg/m²) | Through study completion, average of 18 months
  The BMI is considered one of the parameters regarding obtaining information on the body composition of children
Body fat percentage | Through study completion, average of 18 months
  To assess body fat percentage the results of the BIA, abdominal ultrasound and skinfold measurements will be taken into account
Insulin resistance | Through study completion, average of 18 months
  The assessment of insulin resistance will be made possible through the analysis of the blood sample (glucose and insulin level are measured)
Inflammatory state of the child (hs-CRP and IL-6) | Through study completion, average of 18 months
  The assessment of inflammatory state will be an assessment of the hs-CRP and IL-6 levels taken into account
Lipid state in blood | Through study completion, average of 18 months
  The assessment of lipid state will be an assessment of the total cholesterol, HDL-cholesterol, LDL-cholesterol and triglycerids taken into account

CONTACTS AND LOCATIONS:
Overall Officials: Roland Devlieger, Professor, Study Director — Universitaire Ziekenhuizen KU Leuven; Inge Gies, Professor, Principal Investigator — Universitair Ziekenhuis Brussel; Karolien Van De Maele, M.D., Study Director — Universitair Ziekenhuis Brussel
Locations (1):
- University Hospital of Brussels, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Van De Maele K, Gies I, Devlieger R. Effect of bariatric surgery before pregnancy on the vascular function in the offspring: protocol of a cross-sectional follow-up study. BMJ Paediatr Open. 2019 Jan 31;3(1):e000405. doi: 10.1136/bmjpo-2018-000405. eCollection 2019. PMID 30815589